CLINICAL TRIAL: NCT03244111
Title: Examining the Effect of a Simple Memory Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Daniel Saltel, Community Health Science Msc Student, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2017:105
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Intervention Model Description: The MOCA is a one page test that assesses cognition. The MOCA will be administered and participants with total scores <= 25 will be in the lower cognition group, whereas participants with total scores > 25 will be in the higher cognition group. These are recommended cut off scores to detect mild cognitive impairment (MCI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Cognition (Active Comparator): The intervention will be carried out as described in the study details using the simple memory tool. The group with healthy cognition may perform better on tasks since they have a higher level of cognition.
  Interventions: Behavioral: simple memory tool
- MCI (Active Comparator): The intervention will be carried out as described in the study details using the simple memory tool. The group with MCI may have a lower level of performance on tasks since they have a lower level of cognition. Some tasks may take longer for the participant or need more explanation from the researcher (e.g., explanation of a question).
  Interventions: Behavioral: simple memory tool

INTERVENTIONS:
Behavioral: simple memory tool — The goals may be implemented using the simple memory tool. Simple memory tool involves using materials such as checklists or diaries to assist with memory.

SUMMARY:
Objective: There have been a wide variety of interventions to assist with cognition and memory of older adults; however, it is often unclear if the interventions have an impact on daily life memory performance and goal attainment. The objectives of this study are to examine: 1) whether an intervention that involves a simple memory tool assists with daily life memory performance and goal attainment of older adults; and 2) whether the intervention has a different effect for individuals with healthy cognition versus individuals with mild cognitive impairment (MCI).

Research Questions: Can a simple memory tool assist with daily life memory performance and goal attainment for older adults? Does the simple memory tool have a different effect for individuals with healthy cognition and individuals with MCI? Methods: The study will use a mixed 2 X 3 design with cognition (healthy, MCI) as the between subjects factor and time (session 1, 2, 3) as the within-subjects factor. There will be 40 older adults who have healthy cognition and 20 older adults who have MCI. The study will consist of 3 sessions for each participant. The sessions will be held once a week and incorporate: a) the Montreal Cognitive Assessment (MOCA) to determine level of cognition (healthy, MCI); b) the Prospective and Retrospective Memory Questionnaire (PRMQ) to help determine daily memory performance; c) a memory recall test for recent daily events to help determine daily memory performance; d) the goals of the participants using the Goal Attainment Scaling (GAS); and e) the development of checklists that are tailored to address goals. In between the sessions, participants will perform the checklists and update the diary with notes of what they want to remember on a daily basis. The hypotheses are that: 1) memory performance (i.e., measured with memory recall of daily events and PRMQ), and goal attainment will increase from session to session; 2) participants with healthy cognition will have better memory performance and goal attainment than participants with MCI; and 3) participants with healthy cognition will have greater gains in memory performance and goal attainment than participants with MCI.

DETAILED DESCRIPTION:
Method Participants The sample will consist of older adults (aged 55 or older). There will be 30 participants: 15 participants will have healthy cognition, and 15 participants will have MCI. The sample size was chosen in consideration to assumptions of robustness for repeated measures analysis of variance (ANOVA), and considerations to power (i.e., standard deviation and effect size from the pilot project). Participants will be recruited from the Centre on Aging participant database and the Alzheimer's Society of Manitoba. Individuals who are in the Centre on Aging participant database have given their consent to be contacted by researchers about their willingness to participate in specific research projects. The participants in the database have healthy cognition, and this should provide ample participants for the healthy cognition group for the study. The Centre on Aging participant database has been approved by the Health REB (REB #HS14652). The Alzheimer's Society of Manitoba will be also be contacted to recruit participants because they have contact information of potential participants who have cognitive impairments (i.e., MCI).

Procedure The study will consist of 3 sessions. The sessions will involve a participant meeting with the principal investigator individually for one hour sessions, either at the University of Manitoba (Bannatyne campus or Fort Garry campus), or if participants prefers, in his or her own home.

First session - Preliminary Procedures. During the first session, the principal investigator will describe the project, provide an informed consent form and answer any questions. Once the participant provides written consent, an interview will collect demographics (e.g., age, sex) and memory related information (e.g., difficulties, strategies).

First session - Memory and Goals. Memory assessments will be administered with the MOCA and PRMQ. The researcher will then interview the participant about the participant's memory difficulties and goals the participant has in regards to memory. The interview will be audiotaped and then the goals will be transcribed onto a goals form for the participant's record. A memory recall written test will also be performed that asks participants to list events that they were involved in during the previous week (i.e., the participant's may include events related to goals or any events that they may want to remember).

First session - Work Folder. The researcher and the participant will collaborate to create a daily checklist that the participant will use over the next week. The daily checklist will relate to goals of the participant.

Between Sessions. Between sessions, the participant will use the simple memory tool by using the work materials. The participant will perform tasks from a checklist each day. The participant will also use the pocket notebook to write down any events that they may want to remember (e.g., future tasks that they may want to put on checklists, diary entries that they may later want to transfer to the diary form).

Second Session. The second session will occur 7 days after the first session. Assessments for memory (i.e., memory recall test) and goals (i.e., GAS) will be performed again, similar to the first session. The MOCA will not be needed in the second session since participants have already been assigned to groups (i.e., healthy cognition or MCI). An additional step in the second session will involve goal assessment. The work folder will be updated with updated goals and checklists (i.e., similar to the first session) for the participant to use for the next 7 days.

Third Session. The third session will occur 7 days after the second session. Memory (i.e., PRMQ, memory recall test) and goals (i.e., GAS) will be assessed, similar to the second session. The third session will not include the step for updating work materials with new goals, as this is the last session. An additional step will be to administer a feedback questionnaire to gather feedback and suggestions from the participant on the study.

Tailored Intervention. The checklists are tailored individually to the goals of an individual. Since the intervention has elements that are unique for each individual, an example is included in the appendix to illustrate what the intervention might entail.

ELIGIBILITY:
Inclusion Criteria:

* healthy cognition

  * high level of cognition as determined by MOCA scores
* lower level of cognition as determined by MOCA scores

  * such as mild cognitive impairment (MCI)

Exclusion Criteria:

• If there is impairment that does not allow participants to perform intervention tasks on their own, then assistance may occur by a caregiver. As long as the participant is willing to be involved they can participate in the study. If participants are having too much difficulty they may wish to withdraw from study.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) - Change from baseline to session 2 and 3 | GAS is assessed during session 2 and 3 with the researcher. I.e., Session 1 is the first time the researcher meets with participant, session 2 occurs one week after session 1, session 3 occurs once week after session 2.
  The GAS is a method for measuring goal attainment. It relies on self-report questions that ask if participants met their goals.
Memory Recall Test - Change from sessions 1, 2 and 3 | Memory recall is assessed during session 1, 2 and 3 with the researcher. I.e., Session 1 is the first time the researcher meets with participant, session 2 occurs one week after session 1, session 3 occurs once week after session 2.
  Participants are asked to recall events that occurred last week (i.e., between sessions with the researcher)
Prospective and Retrospective Memory Questionnaire (PRMQ) - Change from session 1 to 3 | PRMQ is assessed during session 1 and 3 with the researcher. I.e., Session 1 is the first time the researcher meets with participant, session 2 occurs one week after session 1, session 3 occurs once week after session 2.
  PRMQ is a questionnaire about daily memory difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Verena Menec, PhD, Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There has been discussion that there may be a follow up study, in which case participant data may be used.